CLINICAL TRIAL: NCT03493451
Title: A Phase 2, Open-Label Study of BGB-A317 in Patients With Relapsed or Refractory Mature T- and NK-cell Neoplasms
Brief Title: Study of BGB-A317 in Participants With Relapsed or Refractory Mature T- and NK-cell Neoplasms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-207; 2017-003700-44 (EudraCT Number); CTR20171387 (Registry Identifier: Center for drug evaluation, CFDA)
Record Dates: First submitted 2018-04-04; First posted 2018-04-10 (Actual); Results first posted 2022-05-04 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Peripheral T Cell Lymphoma; PTCL; Extranodal NK/T-cell Lymphoma; Extranodal NK/T-cell Lymphoma, Nasal Type; Extranodal NK T Cell Lymphoma; Extranodal NK T Cell Lymphoma, Nasal; Adult Nasal Type Extranodal NK/T-cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Angioimmunoblastic T-Cell Lymphoma Recurrent; Angioimmunoblastic T-Cell Lymphoma Refractory; Peripheral T-cell Lymphoma NOS; Peripheral T-Cell Lymphoma, Not Otherwise Specified; Peripheral T-Cell Lymphoma Refractory; Anaplastic Large Cell Lymphoma; Anaplastic Large Cell Lymphoma, ALK-Positive; Anaplastic Large Cell Lymphoma, ALK-negative; ALK-negative Anaplastic Large Cell Lymphoma; ALK-Positive Anaplastic Large Cell Lymphoma; Cutaneous T-cell Lymphoma
Keywords: T/NK-cell; NK/T-cell; extranodal; nasal; NK-cell; ENKTL; peripheral T-cell; anaplastic large cell; ALCL; angioimmunoblastic; PTCL-NOS; Relapsed; Refractory
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, Extranodal NK-T-Cell; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell; Lymphoma, Large-Cell, Anaplastic; Lymphoma, T-Cell, Cutaneous; Recurrence | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: ENKTL (Experimental): Participants with relapsed or refractory (R/R) extranodal natural killer-/T-cell lymphoma (ENKTL; nasal or non-nasal type) were treated with tislelizumab 200 mg intravenously (IV) on Day 1 of each cycle until disease progression, intolerable toxicity, or treatment discontinuation for any other reason (21 days per cycle)
  Interventions: Drug: Tislelizumab
- Cohort 2: PTCL-NOS, AITL, and ALCL (Experimental): Participants with other R/R mature T-cell neoplasms [limited to peripheral T-cell lymphoma-not otherwise specified (PTCL-NOS), angioimmunoblastic T-cell lymphoma (AITL), and anaplastic large-cell lymphoma (ALCL)] were treated with tislelizumab 200 mg intravenously (IV) on Day 1 of each cycle until disease progression, intolerable toxicity, or treatment discontinuation for any other reason (21 days per cycle)
  Interventions: Drug: Tislelizumab
- Cohort 3: MF and SS (Experimental): Participants with R/R cutaneous T-cell lymphoma [limited to mycosis fungoides (MF) and Sèzary syndrome (SS)] were treated with tislelizumab 200 mg intravenously (IV) on Day 1 of each cycle until disease progression, intolerable toxicity, or treatment discontinuation for any other reason (21 days per cycle)
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Administered intravenously
  Other Names: BGB-A317

SUMMARY:
This was a multi-center, prospective, non-randomized, open-label, Phase 2 clinical study to evaluate the safety and efficacy of BGB-A317 in participants with relapsed or refractory mature T- and natural killer (NK)-cell neoplasms. There were three cohorts:

* Cohort 1: Relapsed or refractory (R/R) extranodal NK/T cell lymphoma (ENKTL; nasal or non-nasal type)
* Cohort 2: Other R/R mature T-cell neoplasms, limited to the following histologies: peripheral T-cell lymphoma-not otherwise specified (PTCL-NOS), angioimmunoblastic T-cell lymphoma (AITL), or anaplastic large-cell lymphoma (ALCL)
* Cohort 3: R/R cutaneous T-cell lymphoma, limited to mycosis fungoides (MF) or Sèzary syndrome (SS)

Study procedures included a Screening phase (up to 35 days); Treatment phase (until disease progression, intolerable toxicity, or withdrawal of informed consent, whichever occurs first); Safety Follow-up phase (up to 90 days following last study treatment for all adverse events (AEs) and serious adverse events (SAEs)); and Survival follow-up phase (duration varying by participant).

ELIGIBILITY:
Key Inclusion Criteria

* Confirmed diagnosis of relapsed or refractory extranodal NK/T-cell lymphoma (nasal or non-nasal type, peripheral T-cell lymphoma - not otherwise specified, angioimmunoblastic T-cell lymphoma, anaplastic large cell lymphoma, mycosis fungoides, or Sezary syndrome)
* Age 18 years or older
* Relapsed or refractory to at least 1 prior systemic therapy
* Measurable disease by computed tomography (CT)/magnetic resonance imaging (MRI) for participants in Cohort 1 and 2
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Life expectancy ≥ 6 months
* Adequate respiratory function
* Adequate bone marrow function
* Adequate renal and hepatic function

Key Exclusion Criteria

* Known central nervous system (CNS) involvement by lymphoma
* Previously received immune checkpoint therapy
* Prior malignancy within the past 3 years, except for curatively treated basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast, or localized Gleason score 6 or lower prostate cancer
* Active autoimmune disease or history of autoimmune diseases that may relapse with some exceptions
* Severe or debilitating pulmonary disease
* Clinically significant cardiovascular disease
* Active fungal, bacterial, and/or viral infection requiring systemic therapy
* Known infection with HIV or active viral hepatitis B or C infection
* Major surgery within 4 weeks of the first dose of study drug
* Pregnant or lactating women
* Vaccination with a live vaccine within 35 days prior to the first dose of study drug
* Hypersensitivity to tislelizumab
* Concurrent participation in another therapeutic clinical trial

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (24):
- British Columbia Cancer Agency the Vancouver Centre, Vancouver, British Columbia, Canada
- China (13):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- France (2):
  - Institut Dhematologie de Basse Normandie Chu Caen Normandie, Caen
  - Chu Hopital Lyon Sud, PierreBenite
- Italy (7):
  - Asst Papa Giovanni Xxiii, Medicina Trasfusionale Ed Ematologia, Bergamo
  - Policlinico Sorsola Malpighi, Aou Di Bologna, Bologna
  - Ospedale Policlinico San Martino Irccs Per L Oncologia, Divisione Ematologia Centro Trapianti Di Mid, Genova
  - Ospedale San Raffaele, Milan
  - Ospedale Maggiore, Ematologia E Centro Trapianti Midollo Osseo (Ctmo), Aou Parma, Parma
  - Aou Pisana, Stabilimento Di Santa Chiara, Pisa
  - Azienda Ospedaliera S Maria Di Terni, Terni
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Huiqiang Huang, et al. Tislelizumab (BGB-A317) for relapsed/refractory extranodal NK/T-cell lymphoma: preliminary efficacy and safety results from a phase 2 study. Poster Abstract EP1268, European Hematology Association 2020.
- [Background] Pier Luigi Zinzani, et al. Tislelizumab (BGB-A317) for relapsed/refractory peripheral T-cell lymphomas: Safety and efficacy results from a phase 2 study. Poster Abstract EP1235, European Hematology Association 2020.
- [Derived] Bachy E, Savage KJ, Huang H, Kwong YL, Gritti G, Zhang Q, Liberati AM, Cao J, Yang H, Hao S, Hu J, Zhou K, Petrini M, Russo F, Zhang H, Sang W, Ji J, Ferreri AJM, Damaj GL, Liu H, Zhang W, Ke X, Ghiggi C, Huang S, Li X, Yao H, Paik J, Novotny W, Zhou W, Zhu H, Zinzani PL. Treating relapsed/refractory mature T- and NK-cell neoplasms with tislelizumab: a multicenter open-label phase 2 study. Blood Adv. 2023 Aug 22;7(16):4435-4447. doi: 10.1182/bloodadvances.2022009575. PMID 37276067

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from study centers in Canada, China, France, Italy, and Taiwan, China.
Period: Overall Study
Arm/Group | Cohort 1: ENKTL | Cohort 2: PTCL-NOS, AITL, and ALCL | Cohort 3: MF and SS
Started | 22 | 44 | 11
Completed | 0 | 0 | 0
Not Completed | 22 | 44 | 11
Not completed — Death | 11 | 26 | 3
Not completed — Lost to Follow-up | 1 | 4 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — Progressive Disease | 1 | 0 | 0
Not completed — Transferred to long term extension study | 8 | 13 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: ENKTL | Cohort 2: PTCL-NOS, AITL, and ALCL | Cohort 3: MF and SS | Total
Number analyzed (Participants) | 22 | 44 | 11 | 77
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.5 (16.24) | 55.8 (15.03) | 59.4 (12.45) | 55.1 (15.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 15 | 3 | 26
  Male | 14 | 29 | 8 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 19 | 23 | 2 | 44
  White | 2 | 18 | 8 | 28
  Not Reported | 1 | 3 | 1 | 5
Region of Enrollment [Number; unit: Participants]
  Canada | 0 | 0 | 2 | 2
  China | 19 | 22 | 0 | 41
  Taiwan | 0 | 1 | 0 | 1
  Italy | 2 | 18 | 8 | 28
  France | 1 | 3 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants achieving a best overall response of complete response or partial response as determined by the investigator using Lugano criteria with Lymphoma Response to Immunomodulatory Therapy Criteria (LYRIC) modification for cohorts 1 and 2 and International Society for Cutaneous Lymphomas/European Organization of Research and Treatment of Cancer (ISCL/EORTC) guidelines for cohort 3.
Time Frame: Up to approximately 3 years and 1 week
Population: Safety analysis set includes all participants who received at least one dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: ENKTL | Cohort 2: PTCL-NOS, AITL, and ALCL | Cohort 3: MF and SS
Number analyzed (Participants) | 22 | 44 | 11
Percentage of participants | 31.8 [13.9 to 54.9] | 20.5 [9.8 to 35.3] | 45.5 [16.7 to 76.6]

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR defined as the time from the first determination of an objective response until progression or death, whichever occurs first, as assessed by the investigator using Lugano criteria with LYRIC modification for cohorts 1 and 2 and ISCL/EORTC guidelines for cohort 3.
Time Frame: Up to approximately 3 years and 1 week
Population: Safety analysis set includes all participants who received at least one dose of study drug; Duration of response was summarized for responders (participants who achieved a partial or complete response).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: ENKTL | Cohort 2: PTCL-NOS, AITL, and ALCL | Cohort 3: MF and SS
Number analyzed (Participants) | 7 | 9 | 5
Months | NA [2.66 to NA] — Not estimable due to insufficient number of participants with events (progressive disease or death) | 8.2 [2.50 to NA] — Not estimable due to insufficient number of participants with events (progressive disease or death) | 11.3 [2.76 to 11.30]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from first study drug administration to the date of disease progression or death, whichever occurs first, as assessed by the investigator using Lugano criteria with LYRIC modification for cohorts 1 and 2 and ISCL/EORTC guidelines for cohort 3.
Time Frame: Up to approximately 3 years and 1 week
Population: Safety analysis set includes all participants who received at least one dose of study drug
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: ENKTL | Cohort 2: PTCL-NOS, AITL, and ALCL | Cohort 3: MF and SS
Number analyzed (Participants) | 22 | 44 | 11
Months | 2.7 [1.45 to 5.32] | 2.7 [2.56 to 4.76] | 16.8 [2.60 to 16.82]

4. Secondary Outcome: Overall Survival (OS)
Description: OS defined as the time from first study drug administration to the date of death due to any reason for cohorts 1 and 2.
Time Frame: Up to approximately 3 years and 1 week
Population: Safety analysis set includes all participants who received at least one dose of study drug
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: ENKTL | Cohort 2: PTCL-NOS, AITL, and ALCL
Number analyzed (Participants) | 22 | 44
Months | 8.8 [3.25 to NA] — Upper limit of confidence interval not estimable due to insufficient number of participants with events | 13.3 [7.66 to 26.22]

5. Secondary Outcome: Complete Response Rate (CRR)
Description: CRR is defined as the percentage of participants who achieve complete response or complete metabolic response as best overall response as assessed by the investigator using Lugano criteria with LYRIC modification for cohorts 1 and 2 and ISCL/EORTC guidelines for cohort 3.
Time Frame: Up to approximately 3 years and 1 week
Population: Safety analysis set includes all participants who received at least one dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: ENKTL | Cohort 2: PTCL-NOS, AITL, and ALCL | Cohort 3: MF and SS
Number analyzed (Participants) | 22 | 44 | 11
Percentage of participants | 18.2 [5.2 to 40.3] | 9.1 [2.5 to 21.7] | 9.1 [0.2 to 41.3]

6. Secondary Outcome: Time to Response (TTR)
Description: Time to response defined as the time from first study drug administration to the time the response criteria (complete response or partial response) are first met as assessed by the investigator using Lugano criteria with LYRIC modification for cohorts 1 and 2 and ISCL/EORTC guidelines for cohort 3.
Time Frame: Up to approximately 3 years and 1 week
Population: Safety analysis set includes all participants who received at least one dose of study drug; Time to response was summarized for responders (participants who achieved a partial or complete response).
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1: ENKTL | Cohort 2: PTCL-NOS, AITL, and ALCL | Cohort 3: MF and SS
Number analyzed (Participants) | 7 | 9 | 5
Months | 5.75 [2.1 to 13.9] | 2.86 [2.1 to 5.5] | 6.83 [2.6 to 11.1]

7. Secondary Outcome: Quality of Life Assessment: EQ-5D-5L Change From Baseline in Visual Analogue Score
Description: Mean change from baseline at safety follow-up visit in EQ-5D-5L visual analogue score (VAS). The EQ-5D-5L measures health outcomes using a VAS to record a participant's self-rated health on a scale from 0 to 100, where 100 is 'the best health you can imagine' and 0 is 'the worst health you can imagine.' An increasing score indicates improvements from baseline.
Time Frame: Baseline and on Day 1 in Cycles 5, 9, 13, 17, 21, 25, 29, and 33 (21 days per cycle) and safety follow-up visit (up to 30 days after end of treatment; up to approximately 3 years and 1 week)
Population: Safety analysis set includes all participants who received at least one dose of study drug. The number analyzed represents participants who completed the questionnaire.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: ENKTL | Cohort 2: PTCL-NOS, AITL, and ALCL | Cohort 3: MF and SS
Number analyzed (Participants) | 22 | 44 | 11
Score on a scale
  Cycle 5, Day 1: number analyzed (Participants) | 12 | 19 | 8
  Cycle 5, Day 1 | 4.42 (10.273) | 1.11 (13.884) | 0.25 (22.276)
  Cycle 9, Day 1: number analyzed (Participants) | 6 | 9 | 6
  Cycle 9, Day 1 | 1.17 (4.916) | 5.56 (21.279) | -0.83 (17.713)
  Cycle 13, Day 1: number analyzed (Participants) | 7 | 5 | 6
  Cycle 13, Day 1 | -3.29 (16.650) | 15.00 (19.685) | 1.33 (21.398)
  Cycle 17, Day 1: number analyzed (Participants) | 6 | 6 | 6
  Cycle 17, Day 1 | 0.17 (9.326) | 10.00 (17.889) | 3.67 (23.551)
  Cycle 21, Day 1: number analyzed (Participants) | 4 | 3 | 4
  Cycle 21, Day 1 | 4.25 (10.905) | 8.33 (22.546) | 5.50 (18.285)
  Cycle 25, Day 1: number analyzed (Participants) | 3 | 2 | 2
  Cycle 25, Day 1 | 4.00 (14.422) | -2.50 (10.607) | 5.00 (7.071)
  Cycle 29, Day 1: number analyzed (Participants) | 3 | 2 | 0
  Cycle 29, Day 1 | -2.67 (4.619) | -5.00 (7.071) |
  Cycle 33, Day 1: number analyzed (Participants) | 1 | 1 | 0
  Cycle 33, Day 1 | -3.00 (NA) — Not estimable due to sample size | 0.00 (NA) — Not estimable due to sample size |
  Safety Follow-up: number analyzed (Participants) | 14 | 23 | 2
  Safety Follow-up | -1.50 (8.546) | -9.52 (21.047) | 12.50 (3.536)

8. Secondary Outcome: Quality of Life Assessment: EORTC QLQ-C30 Change From Baseline in Global Health Status Score
Description: Mean change from baseline at safety follow-up visit in EORTC QLQ-C30 Global Health Status/Quality of Life score. The EORTC QLQ-C30 v3.0 is a questionnaire that assesses quality of life of cancer patients and includes global health status and quality of life questions related to their overall health in which participants respond based on a 7-point scale, where 1 is very poor and 7 is excellent. Answers are converted to a score of 0 to 100, with a higher score indicating improved health status.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: ENKTL | Cohort 2: PTCL-NOS, AITL, and ALCL | Cohort 3: MF and SS
Number analyzed (Participants) | 22 | 44 | 11
Score on a scale
  Cycle 5, Day 1: number analyzed (Participants) | 12 | 20 | 8
  Cycle 5, Day 1 | 7.64 (24.220) | 6.67 (19.041) | 10.42 (24.296)
  Cycle 9, Day 1: number analyzed (Participants) | 6 | 9 | 6
  Cycle 9, Day 1 | 8.33 (10.541) | 12.04 (28.294) | 1.39 (21.995)
  Cycle 13, Day 1: number analyzed (Participants) | 7 | 5 | 6
  Cycle 13, Day 1 | 4.76 (11.644) | -1.67 (19.003) | 2.78 (15.516)
  Cycle 17, Day 1: number analyzed (Participants) | 6 | 6 | 6
  Cycle 17, Day 1 | 2.78 (12.546) | 6.94 (30.008) | 4.17 (21.570)
  Cycle 21, Day 1: number analyzed (Participants) | 4 | 3 | 4
  Cycle 21, Day 1 | 12.50 (14.434) | 0.00 (33.333) | 0.00 (20.412)
  Cycle 25, Day 1: number analyzed (Participants) | 4 | 2 | 2
  Cycle 25, Day 1 | 14.58 (25.797) | -8.33 (11.785) | -4.17 (5.893)
  Cycle 29, Day 1: number analyzed (Participants) | 3 | 2 | 0
  Cycle 29, Day 1 | 16.67 (16.667) | -8.33 (11.785) |
  Cycle 33, Day 1: number analyzed (Participants) | 1 | 1 | 0
  Cycle 33, Day 1 | 0.00 (NA) — Not estimable due to sample size | 0.00 (NA) — Not estimable due to sample size |
  Safety Follow-up: number analyzed (Participants) | 14 | 24 | 2
  Safety Follow-up | 7.74 (27.045) | -14.93 (26.917) | 20.83 (17.678)

9. Secondary Outcome: Quality of Life Assessment: EORTC QLQ-C30 Change From Baseline in Fatigue Score
Description: Mean change from baseline at safety follow-up visit in EORTC QLQ-C30 Fatigue score. The EORTC QLQ-C30 v3.0 is a questionnaire that assesses quality of life of cancer patients and includes questions related to fatigue symptoms in which participants respond based on a 7-point scale, where 1 is very poor and 7 is excellent. Answers are converted to a score of 0 to 100, with a higher score indicating improved health status.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: ENKTL | Cohort 2: PTCL-NOS, AITL, and ALCL | Cohort 3: MF and SS
Number analyzed (Participants) | 22 | 44 | 11
Score on a scale
  Cycle 5, Day 1: number analyzed (Participants) | 12 | 19 | 8
  Cycle 5, Day 1 | -2.78 (14.312) | 7.02 (14.912) | 1.39 (41.335)
  Cycle 9, Day 1: number analyzed (Participants) | 6 | 8 | 6
  Cycle 9, Day 1 | 0.00 (12.172) | -1.39 (11.011) | -22.22 (41.574)
  Cycle 13, Day 1: number analyzed (Participants) | 7 | 5 | 6
  Cycle 13, Day 1 | -1.59 (11.878) | -6.67 (12.669) | -5.56 (18.257)
  Cycle 17, Day 1: number analyzed (Participants) | 6 | 6 | 6
  Cycle 17, Day 1 | 9.26 (16.355) | 1.85 (10.924) | -12.96 (16.355)
  Cycle 21, Day 1: number analyzed (Participants) | 4 | 3 | 4
  Cycle 21, Day 1 | 0.00 (12.830) | 11.11 (11.111) | -16.67 (14.344)
  Cycle 25, Day 1: number analyzed (Participants) | 4 | 2 | 2
  Cycle 25, Day 1 | 0.00 (15.713) | 27.78 (7.857) | -5.56 (7.857)
  Cycle 29, Day 1: number analyzed (Participants) | 3 | 2 | 0
  Cycle 29, Day 1 | 3.70 (27.962) | 22.22 (15.713) |
  Cycle 33, Day 1: number analyzed (Participants) | 1 | 1 | 0
  Cycle 33, Day 1 | 11.11 (NA) — Not estimable due to sample size | 33.33 (NA) — Not estimable due to sample size |
  Safety Follow-up: number analyzed (Participants) | 14 | 24 | 2
  Safety Follow-up | -1.59 (19.903) | 7.87 (30.820) | -44.44 (31.427)

10. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), including clinically relevant changes in laboratory tests, physical examination, electrocardiogram, and vital signs
Time Frame: Up to approximately 3 years and 1 week
Population: Safety analysis set includes all participants who received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ENKTL | Cohort 2: PTCL-NOS, AITL, and ALCL | Cohort 3: MF and SS
Number analyzed (Participants) | 22 | 44 | 11
Participants
  At least one TEAE | 22 | 41 | 10
  SAEs | 9 | 21 | 5

ADVERSE EVENTS:
Time Frame: Up to approximately 3 years and 1 week
Description: Adverse events were graded by the investigators using Common Terminology Criteria for Adverse Events (CTCAE) v4.03.
Arm/Group | Cohort 1: ENKTL | Cohort 2: PTCL-NOS, AITL, and ALCL | Cohort 3: MF and SS
All-Cause Mortality (participants affected / at risk) | 11/22 | 26/44 | 3/11
Serious Adverse Events (participants affected / at risk) | 9/22 | 21/44 | 5/11
Other Adverse Events (participants affected / at risk) | 21/22 | 39/44 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: ENKTL (N=22) | Cohort 2: PTCL-NOS, AITL, and ALCL (N=44) | Cohort 3: MF and SS (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (2) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 2 (2) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (3) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 4 (8) | 0 (0)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (5) | 4 (4) | 0 (0)
Pneumonia cryptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Epstein-Barr virus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: ENKTL (N=22) | Cohort 2: PTCL-NOS, AITL, and ALCL (N=44) | Cohort 3: MF and SS (N=11)
Anaemia (Blood and lymphatic system disorders) | 6 (14) | 7 (8) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 5 (13) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 7 (11) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 2 (3) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 5 (5) | 3 (4)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 1 (2)
Eversion of lacrimal punctum (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal disorder (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Retinopathy (Eye disorders) | 3 (3) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 4 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2)
Oral cavity fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (3) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3)
Asthenia (General disorders) | 1 (2) | 8 (9) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (3) | 1 (2)
Influenza like illness (General disorders) | 0 (0) | 1 (2) | 3 (3)
Malaise (General disorders) | 3 (3) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (2)
Oedema peripheral (General disorders) | 2 (2) | 3 (3) | 4 (6)
Pyrexia (General disorders) | 6 (13) | 13 (25) | 4 (7)
Swelling face (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (3) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pseudomonal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Skin bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 5 (8) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (5) | 0 (0)
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 0 (0) | 2 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 3 (3) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 2 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (5) | 1 (2) | 0 (0)
Blood creatine phosphokinase MB increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (5) | 1 (1) | 1 (4)
Blood creatinine increased (Investigations) | 0 (0) | 3 (6) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 4 (7) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (2) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (9) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (16) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 2 (10) | 4 (5) | 0 (0)
Tri-iodothyronine free decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 4 (8) | 4 (5) | 0 (0)
Weight increased (Investigations) | 3 (11) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 4 (21) | 3 (6) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 4 (5) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (8) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (7) | 0 (0) | 0 (0)
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 7 (18) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (4)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 4 (4) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (10) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Circumoral oedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (10) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 6 (9) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 3 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (8) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/51/NCT03493451/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/51/NCT03493451/SAP_001.pdf